CLINICAL TRIAL: NCT04055779
Title: Minimal Inflation Tourniquet Pressure Using Induced Hypotension With Limb Occlusion Pressure Determination or Arterial Occlusion Pressure Estimation in Upper Limb Surgery: A Randomized Double Blinded Comparative Study
Brief Title: Minimal Inflation Tourniquet Pressure Using Induced Hypotension
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Samaa Rashwan, Assistant professor, Beni-Suef University
Other Study IDs: Beni-Suef University Hospital
Record Dates: First submitted 2019-07-27; First posted 2019-08-14 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Vascular Diseases
MeSH Terms: conditions — Vascular Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Induced hypotension and arterial occlusion pressure: The patients will receive induced hypotensive anesthesia and the tourniquet pressure will be based on the the tourniquet pressure will be determined based on the AOP which will be determined by the estimation formula (AOP=[SBP+10]/KTP) . The calculation is based on using initial SBP and tissue padding coefficient values , according to limb circumferences of the patient.After calculation of AOP, tourniquet pressures will be determined by adding a safety margin of 20 mmHg to AOP values(tourniquet pressure=AOP+20 mmHg).
  Interventions: Other: estimation method for arterial occlusion pressure; Other: the limb occlusion pressure
- induced hypotension and limb occlusion pressure: the patients will receive induced hypotensive anesthesia and the tourniquet pressure will be based on the LOP.using the ultrasound Doppler technique and the tourniquet will be inflated until the arterial pulsations disappear at the side of the operation. This pressure will be recorded as LOP .the tourniquet cuff will be inflated to the pressure according to theguidelines of the Association of Perioperative Registered Nurses(AORN) which recommends that a safety margin of 40 mmHg should be added for AOP below 130 mmHg, 60 mmHg for AOP between 131 mmHg and 190 mmHg, and 80 mmHg for AOP above 190 mmHg for adult patients
  Interventions: Other: estimation method for arterial occlusion pressure; Other: the limb occlusion pressure

INTERVENTIONS:
Other: estimation method for arterial occlusion pressure — The patients will receive induced hypotensive anaesthesia and the tourniquet pressure will be based on the AOP.the tourniquet pressure will be determined based on the AOP which will be determined by the estimation formula (AOP=[SBP+10]/KTP) . The calculation is based on using initial SBP and tissue padding coefficient values , according to limb circumferences of the patient.After calculation of AOP, tourniquet pressures will be determined by adding a safety margin of 20 mmHg to AOP values(tourniquet pressure=AOP+20 mmHg).
Other: the limb occlusion pressure — : using the ultrasound Doppler technique and the tourniquet will be inflated until the arterial pulsations disappear at the side of the operation. This pressure will be recorded as LOP.using the ultrasound Doppler technique and the tourniquet will be inflated until the arterial pulsations disappear at the side of the operation. This pressure will be recorded as LOP .the tourniquet cuff will be inflated to the pressure according to theguidelines of the Association of Perioperative Registered Nurses(AORN) which recommends that a safety margin of 40 mmHg should be added for AOP below 130 mmHg, 60 mmHg for AOP between 131 mmHg and 190 mmHg, and 80 mmHg for AOP above 190 mmHg for adult patients

SUMMARY:
Limb occlusion pressure (LOP) and arterial occlusion pressure (AOP) are the terms that mean the lowest tourniquet pressure required to stop the arterial blood flow into the limb distal to the cuff. LOP can be determined manually or automatically by slow cuff inflation until disapper of pulsation with Doppler flow-meter or pulse oximeter

DETAILED DESCRIPTION:
The advantages of the tourniquet during upper or lower limb procedures are providing bloodless operative field and so less intra-operative blood lossIt has been reported that using the lowest effective inflation pressure minimize tourniquet induced nerve injury .). Limb occlusion pressure (LOP) and arterial occlusion pressure (AOP) are the terms that mean the lowest tourniquet pressure required to stop the arterial blood flow into the limb distal to the cuff. LOP can be determined manually or automatically by slow cuff inflation until disapper of pulsation with Doppler flowmeter or pulse oximeter .AOP can be estimated by a formula (AOP = [SBP + 10]/KTP) using patient's systolic blood pressure (SBP) and tissue padding coefficient (KTP) values. In both methods, addition of a safety margin to LOP or AOP is recommended for potential hemodynamic fluctuations during surgery

ELIGIBILITY:
Inclusion Criteria:

* • ASA physical status I and II.

  * Male and female patient
  * Age group 20-50 years old

Exclusion Criteria:

* • Patient who refuse to participate in the study

  * Patients with contraindication of using the tourniquet (e.g. peripheral vascular disease or coronary artery disease sickle cell anemia neuromuscular disorders,)
  * Contraindications of using induced hypotensive anesthesia (cerebrovascular disease, Impaired kidney function , chronic liver disease, pregnancy).
  * Patients on medications inﬂuencing blood ﬂow such as nitrogycerine
  * Surgery extends more than 90 minutes.
  * Hypertensive patients

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study will include the patients scheduled for elective upper limb surgery under general anesthesia who met the inclusion criteria The patient will be scheduled into either group A or B.
  Group (A): The patients will receive induced hypotensive anaesthesia and the tourniquet pressure will be based on the AOP .
  Group (B): the patients will receive induced hypotensive anaesthesia and tourniquet pressure will be based on LOP.
  ,
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2019-11 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Tourniquet inflation pressure | tourniquet inflation pressures will be recorded at 0, 5, 15, 30, 60, and 120 min.
  the tourniquet inflation pressure will be determined based on the Arterial occlusion pressure or the limb occlusion pressure
time required to set the tourniquet inflation pressures | one minute before inflation of the tourniquet cuff
  Time needed to estimate AOP or to determine LOP and set the tourniquet cuff pressure.

SECONDARY OUTCOMES:
tourniquet performance | at the middle and end of surgery
  tourniquet performance as determined by the quality of bloodless surgical field.

CONTACTS AND LOCATIONS:
Overall Officials: Samaa ak Rashwan, MD, Principal Investigator — Assisstant proffesor of anesthesia
Locations (1):
- Beni-Suef University Hospital, Banī Suwayf, Egypt

IPD SHARING:
Plan to Share IPD: No